CLINICAL TRIAL: NCT03209531
Title: Operant Conditioning of Motor Evoked Responses to Improve Quadriceps Function in Individuals With Anterior Cruciate Ligament Reconstruction
Brief Title: Conditioning Brain Responses to Improve Thigh Muscle Function After Anterior Cruciate Ligament Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Medical University of South Carolina (Other); National Center of Neuromodulation for Rehabilitation (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Chandramouli Krishnan, Director of Neuromuscular and Rehabilitation Robotics Laboratory, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00130845; P2CHD086844 (NIH)
Record Dates: First submitted 2017-06-30; First posted 2017-07-06 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Anterior Cruciate Ligament Injury
Keywords: Quadriceps activation deficits; ACL; Surgery; Quadrcieps weakness; Operant conditioning; Cortical excitability
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Operant Conditioning (Experimental): Participants will receive operant conditioning training and single pulse transcranial magnetic stimulation 2-3 times a week for about 8 weeks.
  Interventions: Behavioral: Operant Conditioning; Device: Single Pulse Transcranial Magnetic Stimulation
- Control (Experimental): Participants will receive single pulse transcranial magnetic stimulation 2-3 times a week for about 8 weeks without operant conditioning training.
  Interventions: Behavioral: Control; Device: Single Pulse Transcranial Magnetic Stimulation

INTERVENTIONS:
Behavioral: Operant Conditioning — Active encouragement and feedback to increase motor evoked response when stimulated.
  Arms: Operant Conditioning
Behavioral: Control — Absence of active encouragement and feedback to increase motor evoked response when stimulated.
  Arms: Control
Device: Single Pulse Transcranial Magnetic Stimulation — Transcranial magnetic stimulation to elicit a motor evoked response from the quadriceps muscles.

SUMMARY:
The purpose of this study is to examine if thigh muscle weakness and the lack of muscle activation that accompanies ACL injury can be improved through a form of mental coaching and encouragement, known as operant conditioning.

DETAILED DESCRIPTION:
Thigh muscle weakness is a common result after anterior cruciate ligament (ACL) injury and reconstruction surgery. Therefore, reducing thigh muscle weakness after ACL injury and reconstructive surgery is important as the quadriceps muscles act as shock absorbers that protect the knee joint. If significant weakness is present in the quadriceps, the knee is exposed to increased forces and often results in degeneration of the structures in the joint leading to osteoarthritis. Thus, it is important to investigate activation and strength rehabilitation methods for the quadriceps muscles. This research study is being done to learn if thigh muscle weakness and the lack of muscle activation that accompanies ACL injury can be improved by conditioning brain responses (elicited by non-invasive transcranial magnetic stimulation) using a form of training called as operant conditioning.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-45 years
* suffered an acute, complete ACL rupture
* have undergone ACL reconstructive surgery
* willingness to participate in testing and follow-up as outlined in the protocol

Exclusion Criteria:

* have suffered a previous ACL injury;
* have undergone previous major surgery to either knee;
* have a history of recent significant knee injury (other than ACL) or lower-extremity fracture;
* have a history of uncontrolled diabetes or hypertension;
* be pregnant or plan to become pregnant;
* have metal implants in the head;
* have electronic devices in their ear or heart (e.g., cochlear implants or cardiac pacemakers);
* have unexplained recurrent headaches;
* have a recent history of seizures;
* be taking drugs that reduce seizure threshold;
* have a history of repeated fainting spells;

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2025-11-24 (Actual); Study Completion 2025-11-24 (Actual)

PRIMARY OUTCOMES:
Changes in Quadriceps muscle strength | Approximately 8 weeks after the start of intervention
  Quadriceps strength will be measured using an isokinetic dynamometer. Improvements in quadriceps strength from baseline to the end of intervention will be assessed and compared between groups.

SECONDARY OUTCOMES:
Changes in voluntary activation | Approximately 8 weeks after the start of intervention
  Voluntary activation will be measured using an electrical superimposition technique. Improvements in voluntary activation from baseline to the end of intervention will be assessed and compared between groups.

OTHER OUTCOMES:
Changes in mid-point quadriceps muscle strength | Approximately 4 weeks after the start of intervention (mid-time point evaluation)
  Quadriceps strength will be measured using an isokinetic dynamometer. Improvements in quadriceps strength from baseline to the mid-point of intervention will be assessed and compared between groups.
Changes in mid-point voluntary activation as measured by percentage activation deficit | Approximately 4 weeks after the start of intervention (mid-time point evaluation)
  Voluntary activation will be measured using an electrical superimposition technique. Improvements in voluntary activation from baseline to the mid-point of intervention will be assessed and compared between groups.
Changes in motor cortical excitability measures | Approximately after 8 weeks after the start of intervention
  Motor cortical excitability will be measured using single- and paired-pulse transcranial magnetic stimulation protocols. Improvements in motor cortical excitability from baseline to the end of intervention will be assessed and compared between groups.
Changes in Knee Injury and Osteoarthritis Outcome Score | Approximately after 8 weeks after the start of intervention
  Knee Injury and Osteoarthritis Outcome Score (KOOS) will be measured using the KOOS questionnaire, which is a self-administered survey of knee function across five domains: pain, symptoms, activities of daily living, sport and recreation function, and knee related quality of life (scores range from 0 to 100, with 0 indicating extreme symptoms and 100 indicating no symptoms). The improvements in KOOS from baseline to the end of intervention will be assessed and compared between groups.
Changes in International Knee Documentation Committee Score | Approximately after 8 weeks after the start of intervention
  International Knee Documentation Committee (IKDC) score will be measured using the IKDC subjective knee evaluation form, which is a survey of self-reported level of knee functioning across different domains (scores range from 0 to 100, with 0 indicating extreme symptoms and 100 indicating no symptoms).The improvements in IKDC score from baseline to the end of intervention will be assessed and compared between groups.
Changes in Lysholm Knee Score | Approximately after 8 weeks after the start of intervention
  Lysholm knee score will be measured using the Lysholm Knee Scoring Scale, which is a questionnaire that assesses knee function after conservatively or surgically treated knee ligament injuries based on activities that require knee movement (scores range from 0 to 100, with 0 indicating extreme symptoms and 100 indicating no symptoms). The improvements in Lysholm score from baseline to the end of intervention will be assessed and compared between groups.
Changes in Tegner Activity Score | Approximately after 8 weeks after the start of intervention
  Tegner activity score will be measured using the Tegner Activity level scale, which is a self-reported measure of activity level (scores range from 0 to 10, with 0 indicating no activity because of knee problems and 10 indicating extremely active in competitive sports). The improvements in Tegner activity score from baseline to the end of intervention will be assessed and compared between groups.
Changes in Marx Activity Rating Score | Approximately after 8 weeks after the start of intervention
  Marx activity rating score will be measured using the Marx Activity Rating Scale, which is a self-reported rating scale designed to measure a subject's level of physical activity in four different categories: running, cutting, deceleration and pivoting (scores range from 0 to 16, with 0 indicating very low activity [< one time in a month] because of knee problems and 16 indicating very high activity [> 4 times in a week] in the four categories). The improvements in Marx activity score from baseline to the end of intervention will be assessed and compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Chandramouli Krishnan, PhD, Principal Investigator — Assistant Professor
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States